CLINICAL TRIAL: NCT03268512
Title: The Use of L-PRF and A-PRF in Ridge Preservation: a Randomized Controlled Clinical Trial
Brief Title: Effect of L-PRF and A-PRF in Ridge Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Ana CASTRO SARDA, Doctoral researcher, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B322201525149
Record Dates: First submitted 2017-08-28; First posted 2017-08-31 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Atrophic Maxilla; Ridge Preservation
Keywords: leucocyte- and platelet rich fibrin; ridge preservation; growth factors; platelet concentrates
MeSH Terms: conditions — Atrophic Maxilla

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L-PRF (Experimental): One socket will be filled with L-PRF membranes and covered with at least 2 L-PRF membranes. A modified horizontal mattress will be place as suture to keep the L-PRF in place.
  Interventions: Other: L-PRF
- A-PRF (Experimental): One socket will be filled with A-PRF membranes and covered with at least 2 A-PRF membranes. A modified horizontal mattress will be place as suture to keep the A-PRF in place.
  Interventions: Other: A-PRF
- Control (No Intervention): The socket will be filled with a natural blood clot. A modified horizontal mattress will be place as suture.

INTERVENTIONS:
Other: L-PRF — Platelet concentrates are produced from a small peripheral blood sample, which is immediately centrifuged without any anticoagulant. Coagulation starts during the centrifugation, and three layers are obtained: red blood corpuscles (RBCs) at the bottom of the tube, platelet-poor plasma (PPP) on the top and an intermediate layer called "buffy coat" where most platelets and leucocytes are concentrated. L-PRF has potential advantages, namely: it creates a bioactive construct that stimulates the local environment for differentiation and proliferation of stem and progenitor cells and it acts as an immune regulation node with inflammation control abilities, such as slow continuous release of growth factors over a period of 7-14 days.
  Arms: L-PRF
Other: A-PRF — Platelet concentrates are produced from a small peripheral blood sample, which is immediately centrifuged without any anticoagulant. Coagulation starts during the centrifugation, and three layers are obtained: red blood corpuscles (RBCs) at the bottom of the tube, platelet-poor plasma (PPP) on the top and an intermediate layer called "buffy coat" where most platelets and leucocytes are concentrated. L-PRF has potential advantages, namely: it creates a bioactive construct that stimulates the local environment for differentiation and proliferation of stem and progenitor cells and it acts as an immune regulation node with inflammation control abilities, such as slow continuous release of growth factors over a period of 7-14 days.
  Arms: A-PRF

SUMMARY:
A split-mouth design study will be performed regarding the use of platelet concentrates on ridge preservation: L-PRF vs A-PRF vs control. Patient needing multiple teeth extractions in the upper jaw (single-rooted teeth) will be recruited. The use of each platelet concentrate or control will be randomized by means of a computer program. The results will be analysed clinical and radiographically (CBCT). When the subject will choose for implant rehabilitation, a biopsy will be taken in the site of the preserved sockets. The region will be localized with a customized stent, fabricated with the position of the extracted teeth. VAS scales will be provided to evaluate the post-operative discomfort.

ELIGIBILITY:
Inclusion Criteria:

* 3 single-rooted teeth needed to be extracted in the upper jaw
* patient in good general health as documented by self-assessment
* patients must be committed to the study and must be willing to sing the informed consent.

Exclusion Criteria:

* any systemic medical condition that could interfere with the surgical procedure or planned treatment.
* current pregnancy or breast feeding
* radiotherapy or chemotherapy in head and neck area
* intravenous and oral bisphosphonate
* patients smoking >20 cig/day
* unwillingness to return for the follow-up examination

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08-22 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Changes horizontal width at crest -1mm | 3 months
  Primary outcome variables were deﬁned as the changes in horizontal width at crest-1 mm levels.

SECONDARY OUTCOMES:
Changes horizontal width at crest -3 mm and 5 mm; vertical resorption; socket fill | 3 months
  Changes in horizontal width at crest -3 mm and 5 mm; vertical resorption at the lingual and buccal side; socket ﬁll.

OTHER OUTCOMES:
Post-operative scores | 1 week
  Post-operative discomfort measured with VAS

CONTACTS AND LOCATIONS:
Overall Officials: Ana B Castro, PhD student, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No